CLINICAL TRIAL: NCT00855335
Title: A Single Arm, Open Label Study to Assess the Pharmacokinetics of Darunavir and Ritonavir, Darunavir and Cobicistat, Etravirine, and Rilpivirine in HIV-1 Infected Pregnant Women
Brief Title: A Single-arm, Open-label, Study to Assess the Pharmacokinetics of Darunavir and Ritonavir, Darunavir and Cobicistat, Etravirine, and Rilpivirine in HIV-1 Infected Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015442; TMC114HIV3015 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-05

CONDITIONS: HIV; HIV Infections; Pregnancy
Keywords: HIV-1; HIV; Pregnancy; Postpartum; Human immunodeficiency virus; PREZISTA; INTELENCE; NORVIR; TMC114; TMC125; darunavir; ritonavir; etravirine; rilpivirine; TMC278; Cobicistat; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; etravirine; Rilpivirine; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Darunavir 600 /Ritonavir 100 (Experimental): TMC114 (darunavir) Two 300 milligram (mg) or one 600 mg tablet twice daily up to 12 weeks postpartum / ritonavir one 100 mg tablet twice daily with darunavir up to 12 weeks postpartum.
  Interventions: Drug: Darunavir; Drug: Ritonavir
- Group 2: Darunavir 800/Ritonavir 100 (Experimental): TMC114 (darunavir) 800mg tablet once daily up to 12 weeks postpartum/ ritonavir one 100 mg tablet once daily with darunavir up to 12 weeks postpartum.
  Interventions: Drug: Darunavir; Drug: Ritonavir
- Group 3: Etravirine (Experimental): TMC125 (etravirine) 200 mg (1*200 mg/2*100 mg) tablets twice daily up to 12 weeks postpartum.
  Interventions: Drug: Etravirine
- Group 4: Rilpivirine (Experimental): TMC278 (rilpivirine) One 25 mg tablet once daily up to 12 weeks postpartum.
  Interventions: Drug: Rilpivirine
- Group 5: Darunavir 800/Cobicistat 150 (Experimental): Fixed dose combination (FDC) tablet of TMC114 (darunavir) 800 mg and cobicistat 150 mg once daily up to 12 weeks postpartum.
  Interventions: Drug: Darunavir/Cobicistat (FDC)

INTERVENTIONS:
Drug: Darunavir — TMC114 (darunavir) two 300 mg or one 600 mg tablet twice daily up to 12 weeks postpartum in Group 1. TMC114 (darunavir) 800mg tablet once daily up to 12 weeks postpartum in Group 2.
  Arms: Group 1: Darunavir 600 /Ritonavir 100; Group 2: Darunavir 800/Ritonavir 100
Drug: Ritonavir — 100 mg tablet twice daily up to 12 weeks postpartum.
  Arms: Group 1: Darunavir 600 /Ritonavir 100; Group 2: Darunavir 800/Ritonavir 100
Drug: Etravirine — 200 mg (1*200 mg/2*100 mg) tablets twice daily up to 12 weeks postpartum.
  Arms: Group 3: Etravirine
Drug: Rilpivirine — One 25 mg tablet once daily up to 12 weeks postpartum.
  Arms: Group 4: Rilpivirine
Drug: Darunavir/Cobicistat (FDC) — Fixed dose combination (FDC) tablet of TMC114 (darunavir) 800 mg and cobicistat 150 mg once daily up to 12 weeks postpartum.
  Arms: Group 5: Darunavir 800/Cobicistat 150

SUMMARY:
The purpose of this study is to study how changes in the body during pregnancy influence the blood levels of TMC114 (darunavir) and ritonavir taken together, darunavir and cobicistat taken as a fixed-dose combination, TMC125 (etravirine) taken alone or with darunavir and ritonavir or rilpivirine in patients with human immunodeficiency virus-1 (HIV-1). This study will examine how these drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time. Any pregnant woman who is currently receiving darunavir with ritonavir, darunavir with cobicistat, etravirine or rilpivirine for HIV-1, and who meets the eligibility criteria for the study, will be allowed to enroll. Patients must be willing to remain on study medication during the course of their pregnancy, and 12 weeks postpartum. The information collected may help answer questions about how to best prescribe these three drugs for pregnant women.

DETAILED DESCRIPTION:
There are many biological changes that occur during pregnancy, some of which may affect the way HIV medications are absorbed, distributed and removed within the body. Some medications have been used for HIV treatment during pregnancy, but little is known about how pregnancy affects the class of drugs being used in this study. To participate in this study, patients must be receiving 600mg of TMC114 (darunavir) taken with 100mg ritonavir twice daily or 800mg of TMC114 (darunavir) with 100mg of ritonavir once daily or 800 mg of darunavir taken with 150mg of cobicistat taken once daily or 200mg of TMC125 (etravirine) (with or without darunavir/ ritonavir) taken twice daily or 25mg of TMC278 (rilpivirine) taken once daily plus additional antiretroviral drugs needed to construct an active antiretroviral regimen. Darunavir and ritonavir, darunavir and cobicistat, etravirine, or rilpivirine will be supplied to study participants. Darunavir and ritonavir are human immunodeficiency virus (HIV) protease inhibitors (PIs); cobicistat is a pharmacoenhancer which boosts the levels of darunavir but has no anti-HIV activity; etravirine and rilpivirine are non-nucleoside reverse transcriptase inhibitor (NNRTI) of HIV. Twelve-hour or twenty four-hour blood sampling will be done for each patient at each of three study visits: Visit 4 (2nd trimester), Visit 5 (3rd trimester), and Visit 8 (6-12 weeks postpartum). Eight blood draws will be taken during each visit: One prior to intake of study medication, and one for each of seven post-dose sampling time-points (hours 1, 2, 3, 4, 6, 9 and 12). The study is designed primarily to examine the pharmacokinetics of darunavir/ritonavir (darunavir/r), darunavir/ cobicistat, etravirine or rilpivirine during the second and third trimesters of gestation, as well as postpartum. Pharmacokinetics measures how the body absorbs, distributes and excretes medication. The study will also examine any changes in anti-viral activity during pregnancy, and the postpartum period. It will note any safety and tolerability of the medications used by the mother, and will measure the level of darunavir/ritonavir, darunavir/ cobicistat, etravirine or rilpivirine in the newborn's cord blood at the time of delivery; outcomes for both mother and child will be assessed as well. During the treatment period, patients will be seen at regular visits in the clinic, where the investigator will assess the patient's medical condition, any Adverse Events and study drug compliance. Laboratory evaluations for efficacy and safety will be done at regular visits as well as blood pressure monitoring. Up to forty-eight (48) HIV positive pregnant women will participate in this study. Study enrollment will be closed once 12 evaluable patients taking darunavir/ritonavir once daily, 12 evaluable patients taking darunavir/cobicistat once daily, 12 evaluable patients taking darunavir/ritonavir twice daily, 12 evaluable patients taking etravirine taking twice daily and 12 evaluable patients taking rilpivirine once daily have been enrolled. The study will be conducted at approximately 14 research centers in the United States and 1 in Puerto Rico. In order to participate, patients must be pregnant for 13-24 weeks. The primary purpose (or outcome) of the study is to assess the influence of pregnancy on the pharmacokinetics of darunavir/ritonavir, darunavir/ cobicistat, etravirine or rilpivirine during the second and third trimesters of gestation, as well as postpartum. Darunavir: One 600 mg or two 300 mg tablets taken twice daily by mouth (two or four tablets a day total). Ritonavir: 100mg tablet taken twice daily by mouth (two tablets a day total), together with darunavir. Darunavir: Two 400 mg tablets taken once daily by mouth (two tablets a day total). Ritonavir: 100mg tablet taken once daily by mouth (one tablet a day total), together with darunavir. Darunavir/ cobicistat: a fixed dose combination containing 800mg of darunavir and 150mg of cobicistat. Etravirine: Two 100 mg tablets taken twice daily by mouth (four tablets a day total). Rilpivirine: One 25mg tablet taken once daily by mouth (one tablet a day total). Study medication will be given from the baseline visit (second pregnancy trimester) until Visit 8 (up to 12 weeks after delivery).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females (18-26 weeks of gestation)
* documented HIV-1 infection
* Receiving darunavir/ritonavir, darunavir/cobicistat, etravirine, or rilpivirine at the time of study entry
* Willing to remain on darunavir/ritonavir, darunavir/cobicistat, etravirine, or rilpivirine as well as a background regimen, for the duration of the study, including 12 weeks postpartum
* Able to comply with the protocol requirements and to provide written informed consent.

Exclusion Criteria:

* Patients with any currently active acquired immune deficiency syndrome (AIDS) defining illness and AIDS-related opportunistic infection
* Patients using cytokine inhibitors (e.g., thalidomide), anabolic hormones, cytokines (e.g., IL-2, INF), efavirenz, hydroxyurea, oral hypoglycemics, systemic chemotherapy or known teratogenic agent
* Use of an investigational agent within 90 days
* Any known fetal anomaly
* Any current obstetric complication, including multiple gestations and pre-term labor
* Hepatitis B and/or C virus infection
* Grade 2 or higher anemia
* Thyroid disease
* Uncontrolled Diabetes Mellitus Types I and II, or gestational diabetes, as determined by the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-04-09 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (17):
- United States (16):
  - Daytona Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Port Saint Lucie, Florida
  - West Palm Beach, Florida
  - Savannah, Georgia
  - Chicago, Illinois
  - Springfield, Massachusetts
  - Dearborn, Michigan
  - Syracuse, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Philadelphia, Pennsylvania
  - Bellaire, Texas
- San Juan Pr, Puerto Rico

REFERENCES:
- [Derived] Osiyemi O, Yasin S, Zorrilla C, Bicer C, Hillewaert V, Brown K, Crauwels HM. Pharmacokinetics, Antiviral Activity, and Safety of Rilpivirine in Pregnant Women with HIV-1 Infection: Results of a Phase 3b, Multicenter, Open-Label Study. Infect Dis Ther. 2018 Mar;7(1):147-159. doi: 10.1007/s40121-017-0184-8. Epub 2018 Jan 15. PMID 29335895

RESULTS

PARTICIPANT FLOW:
Groups:
- Darunavir 600 mg /Ritonavir 100 mg Twice Daily: Participants received darunavir 600 milligram (mg) tablets (300*2) and ritonavir 100 mg capsules orally twice daily up to 12 weeks postpartum.
- Darunavir 800 mg /Ritonavir 100 mg Once Daily: Participants received darunavir 800 mg tablets (400*2) and ritonavir 100 mg capsules orally once daily up to 12 weeks postpartum.
- Etravirine 200 mg Twice Daily: Participants received etravirine 200 mg (1*200 mg/2*100 mg) tablets orally twice daily up to 12 weeks postpartum.
- Rilpivirine 25 mg Once Daily: Participants received tablets containing 25 mg rilpivirine (EDURANT or COMPLERA) orally once daily up to 12 weeks postpartum.
- Darunavir 800 mg/Cobicistat 150 mg Once Daily: Participants received darunavir 800 mg and Cobicistat 150 mg in a fixed-dose combination (FDC) as film-coated tablet formulation (PREZCOBIX) orally once daily up to 12 weeks postpartum.
Period: Overall Study
Arm/Group | Darunavir 600 mg /Ritonavir 100 mg Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Started | 18 | 18 | 15 | 19 | 7
Completed | 13 | 16 | 10 | 12 | 6
Not Completed | 5 | 2 | 5 | 7 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 2 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darunavir 600 mg /Ritonavir 100 mg Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily | Total
Number analyzed (Participants) | 18 | 18 | 15 | 19 | 7 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (5.6) | 24.2 (3.45) | 26.3 (4.91) | 27.2 (4.51) | 28.86 (4.71) | 26.1 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 15 | 19 | 7 | 77
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 15 | 19 | 7 | 77

OUTCOME MEASURES:

1. Primary Outcome: Predose (Trough) Plasma Concentration (C0h)
Description: C0h is defined as the predose (trough) plasma concentration or concentration just prior to study drug administration.
Time Frame: Predose on Weeks 24-28 (Visit 4, 2nd trimester), 34-38 (visit 5, 3rd trimester) and 6-12 weeks postpartum (visit 8)
Population: Population analyzed included participants who received at least one dose of study drug with at least one PK blood sample available. Arms were created to report data separately for the treatments and analytes. Here 'N' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily: Participants received darunavir 600 milligram (mg) tablets (300*2) orally twice daily along with ritonavir 100 mg up to 12 weeks postpartum.
- Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily: Participants received ritonavir 100 mg capsules orally twice daily along with darunavir 600 mg tablets up to 12 weeks postpartum.
- Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily: Participants received darunavir 800 mg tablets (400*2) orally once daily along with ritonavir 100 mg up to 12 weeks postpartum.
- Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily: Participants received ritonavir 100 mg capsules orally once daily along with darunavir 800 mg tablets up to 12 weeks postpartum.
- Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily: Participants received darunavir 800 mg along with cobicistat 150 mg in a fixed-dose combination (FDC) as film-coated tablet formulation (PREZCOBIX) orally once daily up to 12 weeks postpartum.
- Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily: Participants received cobicistat 150 mg along with darunavir 800 mg in a fixed-dose combination (FDC) as film-coated tablet formulation (PREZCOBIX) orally once daily up to 12 weeks postpartum.
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 12 | 13 | 17 | 17 | 13 | 15 | 7 | 7
nanogram per milliliter (ng/mL)
  Postpartum (6-12 W): number analyzed (Participants) | 12 | 12 | 16 | 16 | 10 | 11 | 6 | 7
  Postpartum (6-12 W) | 3608 (2812) | 491.4 (472.4) | 2481 (2183) | 147 (198) | 281 (193) | 127 (97.0) | 2811 (2296) | 134 (145)
  2nd Trimester | 2323 (1140) | 225.9 (127.5) | 1793 (964) | 94.2 (102) | 439 (212) | 75.6 (36.2) | 540 (803) | NA (NA) — Here, NA indicates that the data is not reported because the predose plasma concentrations were Below Quantification Limit (BQL) less than (<) 5.00 ng/mL.
  3rd Trimester: number analyzed (Participants) | 12 | 12 | 15 | 15 | 10 | 13 | 6 | 6
  3rd Trimester | 3280 (1466) | 236.0 (108.08) | 1528 (1184) | 74.6 (90.2) | 413 (78.2) | 78.0 (39.1) | 824 (630) | 30.1 (51.5)

2. Primary Outcome: Minimum Plasma Concentration (Cmin)
Description: The Cmin is the minimum observed plasma concentration.
Time Frame: Between Predose and 24 hours postdose at Weeks 24-28 (Visit 4, 2nd trimester), 34-38 (visit 5, 3rd trimester) and 6-12 weeks postpartum (visit 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 12 | 13 | 17 | 17 | 13 | 15 | 7 | 7
nanogram per milliliter (ng/mL)
  Postpartum (6-12 W): number analyzed (Participants) | 12 | 12 | 16 | 16 | 10 | 11 | 6 | 6
  Postpartum (6-12 W) | 2851 (2216) | 264.7 (259.8) | 1473 (1141) | 40.5 (31.4) | 269 (182) | 84.0 (58.8) | 1538 (1344) | 41.4 (49.1)
  2nd Trimester | 1922 (825) | 141.1 (73.78) | 1248 (542) | 32.2 (19.8) | 383 (210) | 54.3 (25.8) | 168 (149) | NA (NA) — Here, NA indicates that the data is not reported because the plasma concentrations were BQL (< 5.00 ng/mL).
  3rd Trimester: number analyzed (Participants) | 12 | 11 | 15 | 15 | 10 | 13 | 6 | 6
  3rd Trimester | 2661 (1269) | 148.1 (52.26) | 1075 (594) | 28.0 (20.5) | 349 (103) | 52.9 (24.4) | 184 (99.0) | NA (NA) — Here, NA indicates that the data is not reported because the plasma concentrations were BQL (< 5.00 ng/mL).

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The Cmax is the maximum observed plasma concentration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 12 | 13 | 17 | 17 | 13 | 15 | 7 | 7
nanogram per milliliter (ng/mL)
  Postpartum (6-12 W): number analyzed (Participants) | 12 | 12 | 16 | 16 | 10 | 11 | 6 | 6
  Postpartum (6-12 W) | 6659 (2364) | 1110 (901.2) | 7310 (1704) | 742 (335) | 569 (261) | 167 (101) | 7918 (2199) | 996 (323)
  2nd Trimester | 4668 (1097) | 546.8 (249.4) | 4964 (1505) | 439 (241) | 774 (300) | 121 (45.9) | 4340 (1616) | 571 (350)
  3rd Trimester: number analyzed (Participants) | 12 | 12 | 15 | 15 | 10 | 13 | 6 | 6
  3rd Trimester | 5328 (1631) | 536.1 (210.6) | 5132 (1198) | 397 (184) | 785 (238) | 123 (47.5) | 4910 (970) | 759 (366)

4. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax)
Description: The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 12 | 13 | 17 | 17 | 13 | 15 | 7 | 7
hour (h)
  Postpartum (6-12 W): number analyzed (Participants) | 12 | 12 | 16 | 16 | 10 | 11 | 6 | 6
  Postpartum (6-12 W) | 3.00 [1.00 to 6.00] | 5.04 [1.02 to 12.08] | 4.00 [1.00 to 6.00] | 4.18 [2.02 to 6.03] | 4.00 [1.00 to 9.00] | 4.00 [2.03 to 25.08] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 4.00]
  2nd Trimester | 3.00 [0.93 to 5.83] | 4.17 [0.93 to 6.08] | 4.00 [3.00 to 6.08] | 5.92 [2.03 to 6.10] | 3.05 [2.00 to 4.00] | 4.00 [1.00 to 9.00] | 4.00 [3.00 to 6.00] | 4.03 [2.00 to 6.00]
  3rd Trimester: number analyzed (Participants) | 12 | 12 | 15 | 15 | 10 | 13 | 6 | 6
  3rd Trimester | 3.00 [1.00 to 11.88] | 4.07 [1.00 to 9.10] | 3.05 [1.00 to 6.00] | 6.00 [2.02 to 6.02] | 3.00 [2.00 to 6.00] | 4.00 [2.00 to 24.93] | 3.50 [2.00 to 6.00] | 3.50 [2.00 to 4.00]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 12 Hours Post-dose (AUC0-12h)
Description: The AUC (0-12) is the area under the plasma concentration-time curve from time zero to 12 hours post dose. The selected arms were based on the dosing frequency (twice daily).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Etravirine 200 mg Twice Daily
Number analyzed (Participants) | 12 | 12 | 13
nanogram*hour per milliliter (ng*h/mL)
  Postpartum (6-12 W): number analyzed (Participants) | 12 | 12 | 10
  Postpartum (6-12 W) | 56890 (26340) | 7406 (6188) | 5004 (2521)
  2nd Trimester: number analyzed (Participants) | 11 | 12 | 13
  2nd Trimester | 39370 (9597) | 3775 (1265) | 6617 (2766)
  3rd Trimester: number analyzed (Participants) | 12 | 12 | 9
  3rd Trimester | 45880 (17360) | 3750 (1336) | 6846 (1482)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 24 Hours Post-dose (AUC0-24h)
Description: The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours post dose. The selected arms were based on the dosing frequency (once daily).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 17 | 17 | 15 | 7 | 7
nanogram*hour per milliliter (ng*h/mL)
  Postpartum (6-12 W): number analyzed (Participants) | 16 | 16 | 11 | 6 | 6
  Postpartum (6-12 W) | 92116 (29241) | 6584 (2861) | 2714 (1535) | 99613 (34862) | 8643 (3187)
  2nd trimester | 62289 (16234) | 3935 (2063) | 1792 (711) | 47293 (19058) | 3862 (2703)
  3rd trimester: number analyzed (Participants) | 15 | 15 | 13 | 6 | 6
  3rd trimester | 61112 (13790) | 3821 (1723) | 1762 (662) | 47991 (9879) | 4736 (2917)

7. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Plasma Viral Load (<) 50 Copies/Milliliter (mL)
Description: Number of participants were assessed with a viral load (VL) lesser than (<) 50 HIV-1 RNA copies/ mL over time.
Time Frame: Up to postpartum (6-12 weeks)
Population: Intent-to-treat (ITT) analysis set is defined as all participants enrolled in this study who took at least one dose of study medication. Here 'N' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Participants
Groups:
- Darunavir 600 mg /Ritonavir 100 Twice Daily: Participants received darunavir 600 milligram (mg) tablets (300*2) and ritonavir 100 mg capsules orally twice daily up to 12 weeks postpartum.
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 16 | 17 | 13 | 19 | 6
Participants
  2nd trimester Less than(<)50 copies/milliLiter(mL) | 6 | 9 | 12 | 13 | 6
  3rd trimester: <50 copies/mL | 5 | 8 | 10 | 13 | 5
  Postpartum (2-5 weeks): <50 copies/mL | 5 | 8 | 9 | 9 | 5
  Postpartum (6-12 weeks): <50 copies/mL | 6 | 7 | 8 | 10 | 5

8. Secondary Outcome: Mean Change From Baseline in Log10 Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Viral Load Value
Description: Mean change from baseline in log 10 HIV-1 RNA VL was assessed up to postpartum (6-12 weeks).
Time Frame: Baseline, 4 weeks after baseline, 2nd and 3rd trimesters of pregnancy and postpartum (2-5 weeks and 6-12 weeks)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Log 10 copies per milliliter (copies/mL)
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 17 | 18 | 15 | 19 | 7
Log 10 copies per milliliter (copies/mL)
  Baseline: number analyzed (Participants) | 17 | 18 | 15 | 19 | 6
  Baseline | 2.12 (0.179) | 1.88 (0.089) | 2.06 (0.206) | 1.84 (0.159) | 1.77 (0.283)
  4 Weeks after Baseline: number analyzed (Participants) | 4 | 10 | 4 | 4 | 0
  4 Weeks after Baseline | -0.26 (0.161) | -0.27 (0.145) | 0.18 (0.182) | 0.20 (0.172) |
  2nd trimester: number analyzed (Participants) | 16 | 17 | 13 | 14 | 7
  2nd trimester | -0.19 (0.106) | -0.16 (0.104) | 0.16 (0.084) | 0.16 (0.074) | 0.1 (0.233)
  3rd trimester: number analyzed (Participants) | 13 | 15 | 11 | 13 | 6
  3rd trimester | -0.31 (0.107) | -0.23 (0.105) | 0.17 (0.105) | 0.25 (0.113) | 0.21 (0.326)
  Postpartum (2-5 weeks): number analyzed (Participants) | 12 | 16 | 11 | 12 | 6
  Postpartum (2-5 weeks) | -0.18 (0.111) | -0.04 (0.146) | 0.13 (0.168) | 0.20 (0.273) | 0.18 (0.304)
  Postpartum (6-12 weeks): number analyzed (Participants) | 13 | 16 | 10 | 12 | 6
  Postpartum (6-12 weeks) | 0.09 (0.268) | 0.11 (0.265) | 0.05 (0.058) | 0.08 (0.138) | 0.23 (0.347)

9. Secondary Outcome: Mean Change From Baseline in CD4+ Cell Count
Description: Mean Change From Baseline in CD4+ Cell Count were assessed for immunology testing.
Time Frame: Baseline, 4 weeks after baseline, 2nd and 3rd trimesters of pregnancy and postpartum (2-5 weeks and 6-12 weeks)
Population: Intent-to-treat (ITT) analysis set is defined as all participants enrolled in this study who took at least one dose of study medication. Here 'N' signified number of participants evaluated for this outcome measure.
Measure: Mean (Standard Error); unit: 10^6 Cells/Liter
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 16 | 18 | 15 | 19 | 7
10^6 Cells/Liter
  Baseline: number analyzed (Participants) | 16 | 18 | 15 | 19 | 6
  Baseline | 466.3 (49.07) | 497.9 (64.60) | 417.47 (80.469) | 495.79 (79.322) | 594.17 (108.151)
  4 Weeks after Baseline: number analyzed (Participants) | 4 | 10 | 4 | 4 | 0
  4 Weeks after Baseline | -14.8 (23.16) | 116.3 (62.41) | 6.25 (26.004) | 24.00 (56.912) |
  2nd trimester: number analyzed (Participants) | 16 | 17 | 13 | 14 | 7
  2nd trimester | 37.1 (23.31) | 154.1 (44.08) | 13.77 (53.225) | 39.21 (36.496) | 13.29 (34.445)
  3rd trimester: number analyzed (Participants) | 13 | 15 | 10 | 13 | 6
  3rd trimester | 83.5 (29.45) | 274.9 (65.41) | 77.30 (30.803) | 89.46 (26.137) | 72.17 (62.882)
  Postpartum (2-5 weeks): number analyzed (Participants) | 10 | 16 | 11 | 12 | 6
  Postpartum (2-5 weeks) | 127.9 (28.53) | 186.0 (43.51) | 115.36 (33.584) | 139.42 (36.972) | 163 (37.177)
  Postpartum (6-12 weeks): number analyzed (Participants) | 13 | 16 | 10 | 11 | 6
  Postpartum (6-12 weeks) | 174.5 (44.98) | 323.0 (63.99) | 154.90 (54.131) | 168.18 (41.345) | 244.67 (100.74)

10. Secondary Outcome: Number of Participants With Resistance at Virological Failure
Description: Resistance analysis was determined using genotypic and phenotypic analysis at the time of virological failure. For participants with a baseline viral load greater than (>) 200 copies/mL, virologic failure was defined as follows: HIV ribonucleic acid (RNA) levels that did not fall by at least 0.5 log 4 weeks after Baseline; viral load >1000 copies/mL (at 2 successive visits) by gestational weeks 34-38; or viral load >200 copies/mL (at 2 successive visits) after reaching a viral load less than or equal to (<=) 200 copies/mL. For participants with a baseline viral load <=200 copies/mL, virologic failure was defined as viral load of >200 copies/mL (at 2 successive visits) at any point during the study.
Time Frame: Up to follow-up phase (16 weeks after postpartum)
Population: Intent-to-treat (ITT) analysis set is defined as all participants enrolled in this study who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 18 | 18 | 15 | 19 | 7
Participants | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Plasma Concentration of Drug in the Cord Plasma and Maternal Plasma Samples Collected at the Time of Delivery
Description: The drug concentrations were evaluated in the cord plasma and maternal plasma samples collected at the time of delivery.
Time Frame: On day of delivery - Intrapartum (Visit 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Darunavir 600 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Ritonavir 100 mg (Darunavir 600/Ritonavir 100 mg) Twice Daily | Darunavir 800 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Ritonavir 100 mg (Darunavir 800/Ritonavir 100 mg) Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg (Darunavir 800/Cobicistat 150 mg) Once Daily | Cobicistat 150 mg (Darunavir 800/Cobicistat 150 mg) Once Daily
Number analyzed (Participants) | 10 | 10 | 16 | 16 | 11 | 9 | 5 | 5
nanogram per milliliter (ng/mL)
  Cord Plasma: number analyzed (Participants) | 10 | 7 | 16 | 16 | 10 | 8 | 5 | 5
  Cord Plasma | 348.4 (322.90) | 17.07 (23.98) | 228 (302) | NA (NA) — The data was not analyzed in case either the cord or maternal plasma concentration was below quantification limit (lesser than (<) 5.00 ng/mL). | 147 (61.3) | 32.8 (16.7) | 125 (106) | NA (NA) — The data was not analyzed in case either the cord or maternal plasma concentration was below quantification limit (lesser than (<) 5.00 ng/mL).
  Maternal Plasma | 2149 (1140) | 316.7 (394.4) | 1663 (1691) | 154 (274) | 421 (157) | 59.0 (34.7) | 857 (885) | 74.5 (109)

12. Secondary Outcome: Number of Infants With Human Immunodeficiency Virus (HIV) Positive Test Result
Description: The infants were evaluated for HIV positive tests using HIV polymerase chain reaction test (PCR).
Time Frame: Birth to age 16 weeks
Population: Infants population whose mothers were included in Intent-to-treat (ITT) analysis set and who were enrolled in this study and took at least one dose of study medication. 'N' signifies number of infants who were born and had HIV test data available.
Measure: Number; unit: infants
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 14 | 17 | 11 | 10 | 6
infants | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to follow up period (16 weeks after postpartum)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Darunavir 600 mg /Ritonavir 100 Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Number analyzed (Participants) | 18 | 18 | 15 | 19 | 7
Participants
  Any AE | 14 | 17 | 12 | 9 | 5
  Any SAE | 6 | 6 | 4 | 4 | 1

ADVERSE EVENTS:
Time Frame: Up to Follow up phase (16 weeks after postpartum)
Description: Intent-to-treat (ITT) analysis set is defined as all participants enrolled in this study who took at least one dose of study medication. The Adverse events were reported as per MedDRA Version 11.1 for darunavir and rilpivirine ; MeDRA version 16.0 for etravirine.
Arm/Group | Darunavir 600 mg /Ritonavir 100 mg Twice Daily | Darunavir 800 mg /Ritonavir 100 mg Once Daily | Etravirine 200 mg Twice Daily | Rilpivirine 25 mg Once Daily | Darunavir 800 mg/Cobicistat 150 mg Once Daily
Serious Adverse Events (participants affected / at risk) | 6/18 | 6/18 | 4/15 | 4/19 | 1/7
Other Adverse Events (participants affected / at risk) | 13/18 | 17/18 | 12/15 | 8/19 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir 600 mg /Ritonavir 100 mg Twice Daily (N=18) | Darunavir 800 mg /Ritonavir 100 mg Once Daily (N=18) | Etravirine 200 mg Twice Daily (N=15) | Rilpivirine 25 mg Once Daily (N=19) | Darunavir 800 mg/Cobicistat 150 mg Once Daily (N=7)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Medical Observation (Investigations) | 1 | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Gestational Diabetes (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 0
Intra-Uterine Death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 1 | 0
Pregnancy Induced Hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 1 | 0
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir 600 mg /Ritonavir 100 mg Twice Daily (N=18) | Darunavir 800 mg /Ritonavir 100 mg Once Daily (N=18) | Etravirine 200 mg Twice Daily (N=15) | Rilpivirine 25 mg Once Daily (N=19) | Darunavir 800 mg/Cobicistat 150 mg Once Daily (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1 | 1 | 1
Anaemia of Pregnancy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 0
Influenza Like Illness (General disorders) | 2 | 1 | 0 | 0 | 0
Pitting Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Genital Herpes (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea Pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0
Vaginal Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Vaginitis Bacterial (Infections and infestations) | 2 | 2 | 1 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Eye Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Albumin Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Amylase Increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Methicillin-Resistant Staphylococcal Aureus Test Positive (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Streptococcal Identification Test Positive (Investigations) | 0 | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gestational Diabetes (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 2 | 0 | 1
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Labour Pain (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Pregnancy Induced Hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1 | 0
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 4 | 2 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Postpartum Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Genital Discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 0 | 1
High Density Lipoprotein Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine with Aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Poor Quality Sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Uterine Contractions During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pelvic Discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.